CLINICAL TRIAL: NCT02852512
Title: Perspective Randomized Trial Comparing Laparoscopic Vs Robotic-assisted Colposacropexy for Pelvic Organ Prolapse Repair
Brief Title: Trial Comparing Laparoscopic Vs Robotic-assisted Colposacropexy for Pelvic Organ Prolapse Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Elisabetta Costantini, associate professor, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LVR1
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: Laparoscopic Sacrocolpopexy; Robotic Assisted Sacrocolpopexy; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic sacrocolpopexy (Active Comparator): The surgical technique will be the same between the two approaches, in this arm the approach will be laparoscopic
  Interventions: Procedure: sacrocolpopexy
- Robotic assisted Sacrocolpopexy (Active Comparator): The surgical technique will be the same between the two approaches, in this arm the approach will be robotic assisted
  Interventions: Procedure: sacrocolpopexy

INTERVENTIONS:
Procedure: sacrocolpopexy — Peritoneal incision from the sacral promontory to the Pouch of Douglas. After careful dissection of the inter-rectovaginal space, a two-piece Y-shaped polypropylene mesh was fixed posteriorly to the levator ani muscles using a absorbable suture. The midpoint of the mesh is anchored to the posterior wall of the vagina. The anterior portion of mesh was then introduced and fixed within the intervesico- vaginal space to the anterior/apical vaginal wall with a running suture. The tails of both meshes were fixed to the sacral promontory with a strong non-absorbable polypropylene suture. The peritoneal incision was re- approximated with a running absorbable suture

SUMMARY:
The aim of the study is to perspectively compare the anatomical and functional outcomes of Pelvic Organ Prolapse (POP) repair after Laparoscopic or Robotic-assisted Colposacropexy.

DETAILED DESCRIPTION:
Female pelvic floor disorders rank amongst the most common disorders affecting women and include conditions such as urinary incontinence and pelvic organ prolapse (POP). POP is estimated to affect 30% of women aged 50- 89 years, and the lifetime risk of requiring surgery is 11%. Open abdominal sacrocolpopexy is the established gold standard procedure and is indicated when there is prolapse of the anterior and/or apical vaginal wall compartments. Laparoscopic sacrocolpopexy (LSCP) has not been widely adopted as it demands skill and motivation and it is associated with a long learning curve. So the hypothesis is that robot-assisted laparoscopic approach for sacrocolpopexy (RALSCP) could be an alternative to a pure laparoscopic technique.

In the study design 62 patients will be randomly enrolled (31 in the laparoscopic arm and 31 in the robotic assisted one). The primary outcome will be the anatomic one, secondary outcomes will be functional in terms of storage or voiding dysfunctions, sexual dysfunctions, bowel dysfunctions, QoL, post operative complications.

For continuous variables will be used the Mann-Withney test, for categorical data will be used McNemar test and X2 test.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic POP >2 stage according to POP Q system

Exclusion Criteria:

* Obesity
* Heart failure (NYHA III-IV)
* High stage COPD (Chronic Obstructive Pulmonary Disease)
* Patients who underwent more than 2 previous abdominal surgical procedures

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Anatomical outcome | 12 months
  POP <2 according to POP-Q system

SECONDARY OUTCOMES:
Intraoperative ando post operative complications | during surgery and within 90 days after surgery
  Clavien-Dindo classification of surgery complications
post operative pain | within 7 days after surgery
  VAS score (Visual Analog Pain Scale)
voiding and storage symptoms | 2, 6, 12 months after surgery
  fill in Urinary Distress Inventory short form (UDI-6) to assess urinary symptoms
sexual dysfunctions | 2, 6, 12 months after surgery
  fill in Female Sexual Function Index questionnaire (FSFI)
patient satisfaction | 12 months after surgery
  fill in Patient Global Impression of Improvement (PGI-I)
Quality of life | 2, 6, 12 months
  fill in Incontinence Impact Questionnaire-Short form (IIQ-7)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Costantini, MD, Principal Investigator — University Of Perugia
Locations (1):
- Santa Maria della Misericordia Hospital- University of Perugia, Perugia, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee RK, Mottrie A, Payne CK, Waltregny D. A review of the current status of laparoscopic and robot-assisted sacrocolpopexy for pelvic organ prolapse. Eur Urol. 2014 Jun;65(6):1128-37. doi: 10.1016/j.eururo.2013.12.064. Epub 2014 Jan 8. PMID 24433811
- [Result] Seror J, Yates DR, Seringe E, Vaessen C, Bitker MO, Chartier-Kastler E, Roupret M. Prospective comparison of short-term functional outcomes obtained after pure laparoscopic and robot-assisted laparoscopic sacrocolpopexy. World J Urol. 2012 Jun;30(3):393-8. doi: 10.1007/s00345-011-0748-2. Epub 2011 Aug 20. PMID 21858540
- [Result] Awad N, Mustafa S, Amit A, Deutsch M, Eldor-Itskovitz J, Lowenstein L. Implementation of a new procedure: laparoscopic versus robotic sacrocolpopexy. Arch Gynecol Obstet. 2013 Jun;287(6):1181-6. doi: 10.1007/s00404-012-2691-x. Epub 2012 Dec 30. PMID 23274792